CLINICAL TRIAL: NCT01928108
Title: Do Different Methods of Educating Patients Regarding Fluid Intake Reduce Kidney Stone Risks?
Brief Title: Fluid Intake Application to Reduce Kidney Stone Risks
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: 13-2453
Record Dates: First submitted 2013-08-20; First posted 2013-08-23 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Kidney Stone
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- iPhone Application: Participants using an iPhone will download the "waterlogged" application and use this to track daily water intake for 1 week.
  Interventions: Behavioral: iPhone Application
- Android Application: Participants using an Android cell phone will download the "water your body" application and use this to track daily water intake for 1 week.
  Interventions: Behavioral: Android Application

INTERVENTIONS:
Behavioral: iPhone Application — The iPhone application "waterlogged" will be used by participants using and iPhone cellular device. This application will be used to track daily fluid intake for 1 week.
  Groups: iPhone Application
Behavioral: Android Application — The Android application "water my body" will be used by participants using an Android cellular device. This application will be used to track daily fluid intake for 1 week.
  Groups: Android Application

SUMMARY:
The purpose of this investigation is to prospectively evaluate the benefit of different methods of educating patients regarding their fluid intake through a readily available daily cellular phone application to improve overall urine output and reduce risk factors for stone recurrence.

DETAILED DESCRIPTION:
The prevalence of kidney stone disease in the United States is increasing. Recurrence of kidney stone disease has been reported as high as 50% at five years. Urine supersaturation is a predominant factor in the formation of crystallization and stone disease and is dependent on fluid volume. High fluid consumption that dilutes the urine has been shown both in vitro and in clinical studies to reduce the tendency for stone crystallization as well as effectively decrease stone recurrence. As a result, water intake greater than two liters per day is a common initial therapy for prevention of stone disease. However, studies have shown that despite physician counseling most patients are only able to modestly increase their urine volume through fluid intake. This finding may be due to a discrepancy in patient perception of their actual fluid intake and resulting urine volume. The purpose of this investigation is to prospectively evaluate the benefit of different methods of educating patient regarding their fluid intake through a readily available daily cellular phone application to improve overall urine output and reduce risk factors for stone recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years old
2. Seen in urology or nephrology clinic at UNC with a diagnosis of kidney stone
3. Prior 24-hour urine result with volume less than 2 to 2.5 liters

Exclusion Criteria:

1. Patient without cellular phone capable of utilizing Android / Apple application
2. Patient already using some form of monitoring fluid intake / volume
3. Inability to take fluid by mouth
4. Patient with urinary diversion, chronic diarrhea, bowel diversion or other forms of excessive fluid loss
5. Inability to obtain informed consent
6. Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be Patients ≥ 18 years old, seen in urology or nephrology clinic with a diagnosis of kidney stone, and had a prior 24-hour urine result with volume less than 2 to 2.5 liters
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-07; Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-16 (Actual)

PRIMARY OUTCOMES:
24-hour urine volume | 7-10 days from baseline

SECONDARY OUTCOMES:
Actual 24-hour urine volume vs. patient perceived urine volume | 7-10 days from baseline
Ease and interest in monitoring fluid intake based on survey data | 7-10 days from baseline

OTHER OUTCOMES:
24-hour urine volume for study participants vs. urine volume for retrospective cohort of previously treated kidney stone patients | 7-10 days from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Davis Viprakasit, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- North Carolina Memorial Hospital, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Scales CD Jr, Smith AC, Hanley JM, Saigal CS; Urologic Diseases in America Project. Prevalence of kidney stones in the United States. Eur Urol. 2012 Jul;62(1):160-5. doi: 10.1016/j.eururo.2012.03.052. Epub 2012 Mar 31. PMID 22498635
- [Background] Preminger GM. Renal calculi: pathogenesis, diagnosis, and medical therapy. Semin Nephrol. 1992 Mar;12(2):200-16. PMID 1561497
- [Background] Pak CY, Sakhaee K, Crowther C, Brinkley L. Evidence justifying a high fluid intake in treatment of nephrolithiasis. Ann Intern Med. 1980 Jul;93(1):36-9. doi: 10.7326/0003-4819-93-1-36. PMID 7396311
- [Background] Borghi L, Meschi T, Amato F, Briganti A, Novarini A, Giannini A. Urinary volume, water and recurrences in idiopathic calcium nephrolithiasis: a 5-year randomized prospective study. J Urol. 1996 Mar;155(3):839-43. PMID 8583588
- [Background] Parks JH, Goldfischer ER, Coe FL. Changes in urine volume accomplished by physicians treating nephrolithiasis. J Urol. 2003 Mar;169(3):863-6. doi: 10.1097/01.ju.0000044922.22478.32. PMID 12576800